CLINICAL TRIAL: NCT05984914
Title: Psychological and Biological Outcomes in Breast Cancer Patients After Pythagorean Self-Awareness Intervention.
Brief Title: Stress Management and Biological Age in Breast Cancer Patients.RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Charalampopoulou (Other)
Collaborators: Hippocration General Hospital (Other); Saint Savvas Anticancer Hospital (Other); Hellenic Anticancer Institute (Unknown)
Responsible Party: Sponsor-Investigator, Maria Charalampopoulou, PhD candidate, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2513
Record Dates: First submitted 2023-07-23; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Stress; Breast Cancer; Telomere Length, Mean Leukocyte
Keywords: Stress; Breast Cancer; Lifestyle; Stress management; Telomeres; Biological age; PSAI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSAI group (Experimental): Participants are enrolled in the Pythagorean Self-Awareness Intervention (PSAI) where they receive weekly group sessions of 120 min for 8 weeks and they receive information about stress and lifestyle modifications and they are also instructed to practice the PSAI at bedtime and in the morning, every day, at home.
  Interventions: Behavioral: PSAI
- Control group (Active Comparator): One day seminar where they receive information about stress and lifestyle modifications
  Interventions: Behavioral: One day seminar

INTERVENTIONS:
Behavioral: PSAI — The 8 sessions included biofeedback training in diaphragmatic breathing, information about distress, its symptoms, ways to manage stress through lifestyle modifications (physical activity, principals of Mediterranean diet without alcohol consumption, sleep hygiene, diaphragmatic breathing, conflict avoidance) & instructions for lymphedema prevention, introduction to the Pythagorean Self-Awareness Intervention, instructions for the implementation of the technique, analysis of the Golden Verses,and their connection with lifestyle medicine as well as active involvement of the participants with group conversation and sharing of experiences.
  Other Names: Pythagorean Self-Awareness Intervention
  Arms: PSAI group
Behavioral: One day seminar — The one day seminar included biofeedback training in diaphragmatic breathing, information about distress, its symptoms, ways to manage stress through lifestyle modifications (physical activity, principals of Mediterranean diet without alcohol consumption, sleep hygiene, diaphragmatic breathing, conflict avoidance) & instructions for lymphedema prevention.
  Arms: Control group

SUMMARY:
Intense stress has harmful effects on the body, contributing to various disorders. Breast cancer patients experience a build-up of stress due to their diagnosis and treatments. Stress can cause epigenetic changes in a cellular level (such as accelerated increase in biological age) that may negatively affect oncological treatments.

This study aims to investigate the effect of stress management, specifically the Pythagorean Self-Awareness Intervention, on telomere length in T-leukocytes of breast cancer patients after completing all treatments except hormonal therapy. The study involves self-referred questionnaires, hair cortisol collection, and blood material extraction.

Understanding the role of stress management in breast cancer may lead to improved patient outcomes and survival rates.

DETAILED DESCRIPTION:
Distress can have serious effects on the human body and is known to contribute to various disorders, including cardiovascular diseases. In the case of breast cancer, patients often experience a build-up of stressful events throughout their journey with the disease, such as diagnosis, surgery, chemotherapy, radiotherapy, survival, and dealing with side effects of anticancer therapy.

Many studies have shown that psychological stress is closely related to increased cortisol levels in the body. This stress may lead to epigenetic changes in telomere length, the action of telomerase, the function of T-leukocytes, and the response of pro-inflammatory cytokines, all of which play significant roles in the treatment of oncological patients.

Considering these factors, managing stress becomes crucial, as it can not only indirectly affect the disease's outcome but also impact survival. This scientific protocol aims to investigate the impact of a holistic stress management program on the telomere length of T-leukocytes in the peripheral blood of women diagnosed with breast cancer.

The stress management technique to be employed is the Pythagorean Self-Awareness Intervention, which will be administered only after completing all cancer treatments, except for hormonal therapy. The methods that will be followed include distributing self-referred questionnaires to assess stress and lifestyle, collecting hair cortisol samples, and extracting genetic (DNA) material to study the telomere length of T-cells from peripheral blood.

By studying the impact of stress and its management on telomere length in breast cancer patients, this study aims to contribute to a better understanding of how stress affects health outcomes and potentially provide insights into improving patient care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary breast cancer
* Completion of anticancer therapy (except for hormonal therapy)

Exclusion Criteria:

* Psychiatric diagnosis and treatment
* Metastasis
* Previous participation in any stress management and health promotion study
* Inability to read or write in Greek

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Psychological I | 9 weeks after the 1st session
  Perceived stress (measured by Perceived Stress Scale-14, expected decrease in mean score)
Psychological II | 9 weeks after the 1st session
  Symptoms of anxiety-stress-depression (measured by Depression Anxiety Stress Scale-21, expected decrease in mean scores)
Physical I | 9 weeks after the 1st session
  Telomere length (measured in mean T/S)
Physical II | 9 weeks after the 1st session
  Hair cortisol levels (measured in pg/mg )

SECONDARY OUTCOMES:
Physical III | 9 weeks after the 1st session
  Body Composition Analysis (measured in kg and %)
Psychological III | 9 weeks after the 1st session
  QOL (measured by European Organization for Research and Treatment Questionnaire, expected increase in means score)

CONTACTS AND LOCATIONS:
Overall Officials: Flora Bacopoulou, MD,PhD, Study Director — Aghia Sofia Hospital
Locations (1):
- Agios Savvas Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study
Access Criteria: On request

REFERENCES:
- [Background] Chrousos GP. Stress and disorders of the stress system. Nat Rev Endocrinol. 2009 Jul;5(7):374-81. doi: 10.1038/nrendo.2009.106. Epub 2009 Jun 2. PMID 19488073
- [Background] Lin Y, Wang C, Zhong Y, Huang X, Peng L, Shan G, Wang K, Sun Q. Striking life events associated with primary breast cancer susceptibility in women: a meta-analysis study. J Exp Clin Cancer Res. 2013 Aug 13;32(1):53. doi: 10.1186/1756-9966-32-53. PMID 23941600
- [Background] Damjanovic AK, Yang Y, Glaser R, Kiecolt-Glaser JK, Nguyen H, Laskowski B, Zou Y, Beversdorf DQ, Weng NP. Accelerated telomere erosion is associated with a declining immune function of caregivers of Alzheimer's disease patients. J Immunol. 2007 Sep 15;179(6):4249-54. doi: 10.4049/jimmunol.179.6.4249. PMID 17785865
- [Background] Charalampopoulou M, Bacopoulou F, Syrigos KN, Filopoulos E, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on breast cancer patients undergoing adjuvant therapy: A pilot randomized controlled trial. Breast. 2020 Feb;49:210-218. doi: 10.1016/j.breast.2019.12.012. Epub 2019 Dec 20. PMID 31901782
- [Background] Carlson LE, Beattie TL, Giese-Davis J, Faris P, Tamagawa R, Fick LJ, Degelman ES, Speca M. Mindfulness-based cancer recovery and supportive-expressive therapy maintain telomere length relative to controls in distressed breast cancer survivors. Cancer. 2015 Feb 1;121(3):476-84. doi: 10.1002/cncr.29063. Epub 2014 Nov 3. PMID 25367403